CLINICAL TRIAL: NCT01134068
Title: Age-adjusted D-dimer Cut-off Levels to Rule Out Pulmonary Embolism: a Prospective Outcome Study.
Brief Title: Age-adjusted D-dimer Cut-off Levels to Rule Out Pulmonary Embolism
Acronym: ADJUST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marc Righini (Other)
Collaborators: University Hospital, Brest (Other); University Hospital, Angers (Other Government); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor-Investigator, Marc Righini, MD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ADJUST
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2013-04

CONDITIONS: Pulmonary Embolism
Keywords: D-dimer; Pulmonary embolism; Diagnostic strategy; Safety of ruling PE with and age-adjusted DD cut-off
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Evaluation of a modified DD cut-off to rule out PE — Evaluation of a modified DD cut-off to rule out PE

SUMMARY:
Suspected pulmonary embolism (PE) is a frequent clinical problem and remains a diagnostic challenge. The diagnostic approach of PE relies on sequential diagnostic tests, such as plasma D-dimer measurement, multi-slice computed tomography (MSCT) and pulmonary angiography. In addition, the diagnostic workup is usually stratified according to the clinical probability of pulmonary embolism. Clinical probability has a fair predictive accuracy either evaluated implicitly or by clinical prediction rules1 and is useful for identifying patients with a low prevalence of pulmonary embolism who can be usually fully investigated by non invasive tests.The D-dimer test has been extensively evaluated in the exclusion of pulmonary embolism, particularly in outpatients. ELISA D-dimer and second-generation latex agglutination (immuno-turbidimetric tests) have a remarkably high sensitivity and have been proved safe first-line tests in association with clinical probability to rule out pulmonary embolism in outcome studies. The clinical usefulness of D-dimer is defined by the proportion of patients in whom pulmonary embolism may be ruled out by a normal result and it is determined by the specificity. However, ELISA and second-generation latex agglutination (immuno-turbidimetric tests) tests have a quite limited overall specificity of around 35% to 40%. Therefore, many investigators tried to increase the D-dimer thresholds in particular in elderly patients to increase the rate of patients in whom the diagnosis could be excluded by this easy and inexpensive test. Several studies have shown that D-dimer levels increase with age and which turns in a decreased specificity of the D-dimer test at the usual threshold in the elderly, and thus to a less useful test to exclude PE in older patients. Indeed, ELISA D-dimer is able to rule out PE in 60% of patients aged less than 40 years, but in only 5% of patients above the age of 80.8 In this study, raising the cut-off value to various points between 600 ng/ml and 1000 ng/ml increased specificity, but this came at the cost of safety with more false negative test results. In this analysis, however, no stratification was made for clinical probability and the sample was small.

Recently, the investigators retrospectively assessed the value of a progressive cut-off adjusted to age in a wide sample of 1712 patients. This "new" cut-off was defined for D-Dimer test positivity in each patient by multiplying patient's age by 10. All patients with a D-Dimer level below 500mg/ml, and all patients above 50 years whose D-Dimer levels were inferior to their age multiplied by 10 were considered as having a negative D-Dimer test. The exact derivation and validation of this "new" D-dimer cut-off is described hereafter. Using the conventional cutoff, the VIDAS® D-Dimer test was negative (below 500 mg/ml) in 512/1712 patients (29.9%) and none had PE during initial workup or the three-month follow-up period.

Using the cutoff adjusted to age (cutoff for D-Dimer test positivity equals age multiplied by ten, in mg/ml), the figure was as follows. D-Dimer levels were below the adjusted cutoff in 615/1712 patients (35.9%, number needed to test 2.8). This represented a statistically significant 20.1% increase in the number of patients in whom the D-Dimer test was considered as negative, p=0.0002. Of these 615 patients, 5 had PE during initial workup (0.8%, 95 percent confidence interval 0.4 to 1.9%).

These data suggest that adopting this progressive cut-off in patients above 50 years, could increase of about 20% the number of patients in whom PE could be excluded without further testing, with an acceptable safety profile as the three-month thromboembolic rate remained very low.

Therefore, the investigators plan a prospective outcome study in which this progressive or "new" cut-off (age X 10 ng/ml) in patients above 50 years will be used. In this multicentre study, clinical probability will be assessed by the simplified revised Geneva revised score (Table 1) and an ELISA D-dimer test will be performed [Vidas D-Dimer Exclusion® test (Biomérieux, Marcy l'Etoile, Paris, France)]. Patients with a non high clinical probability with the simplified revised Geneva score and a normal "new" D-dimer cut-off with the Vidas D-dimer Exclusion®, (Biomerieux, Marcy l'Etoile, France) will be considered as not having PE, and will be followed for three-months to assess possible VTE recurrences. The main outcome will be the rate of thromboembolic events during a formal 3-month follow-up in patients not anticoagulated on the basis of this strategy. Patients with positive D-dimers will be investigated with MSCT as currently admitted.

ELIGIBILITY:
Inclusion Criteria:

All outpatients admitted to the emergency ward for suspected pulmonary embolism defined as acute onset of new or worsening shortness of breath or chest pain without another obvious etiology will be included in the study, provided they correspond to the following diagnostic and exclusion criteria and they have signed an informed consent form.

Exclusion Criteria:

* PE suspicion raised more than 24 hours after admission to the hospital
* Absence of informed consent
* Incapacity to deliver informed consent
* Life expectancy less than 3 months
* Geographic inaccessibility for follow-up
* Pregnancy.
* Patients anticoagulated for a disease other than venous thromboembolism (for instance, atrial fibrillation)
* Patients allergic to contrast medium
* Impaired renal function (creatine clearance less than 30 ml/min as calculated by the Cockroft formula).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3306 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The main outcome is the rate of thromboembolic events during a formal 3-month follow-up in patients not anticoagulated on the basis of a PE ruled out by the association mentioned here above. | 3 months

SECONDARY OUTCOMES:
Prospective validation of the simplified revised Geneva score. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc Righini, MD, Principal Investigator — University Hospital, Geneva; Grégoire Le Gal, Prof, Principal Investigator — University Hospital, Brest; Renée Douma, MD, Principal Investigator — Amsterdam University Hospital; Pierre-Marie Roy, Prof, Principal Investigator — Angers University Hospital
Locations (4):
- France (2):
  - Grégoire Le Gal, Brest, Brest
  - Angers University Hospital, Angers, France
- Amsterdam University hospital, Amsterdam, Amsterdam, Netherlands
- Geneva University Hospital, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Righini M, Van Es J, Den Exter PL, Roy PM, Verschuren F, Ghuysen A, Rutschmann OT, Sanchez O, Jaffrelot M, Trinh-Duc A, Le Gall C, Moustafa F, Principe A, Van Houten AA, Ten Wolde M, Douma RA, Hazelaar G, Erkens PM, Van Kralingen KW, Grootenboers MJ, Durian MF, Cheung YW, Meyer G, Bounameaux H, Huisman MV, Kamphuisen PW, Le Gal G. Age-adjusted D-dimer cutoff levels to rule out pulmonary embolism: the ADJUST-PE study. JAMA. 2014 Mar 19;311(11):1117-24. doi: 10.1001/jama.2014.2135. PMID 24643601